CLINICAL TRIAL: NCT06633718
Title: A Phase 3,Multicenter, Randomized, Double-Blind, Positive Control，Study to Assess the Efficacy and Safety of Meropenem and Pralurbactam in Complicated Intra-abdominal Infections
Brief Title: Study to Assess the Efficacy and Safety of Meropenem and Pralurbactam in CIAI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FL058-301
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Intra-abdominal Infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — Meropenem; Sodium Chloride; avibactam, ceftazidime drug combination; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem and Pralurbactam (Experimental): Meropenem and Pralurbactam (120min infusion)
  Interventions: Drug: Meropenem and Pralurbactam; Drug: Saline
- Ceftazidime-avibactam (Active Comparator): Ceftazidime-avibactam (120min infusion) 、 Metronidazole(60min infusion)
  Interventions: Drug: Ceftazidime-avibactam; Drug: Metronidazole

INTERVENTIONS:
Drug: Meropenem and Pralurbactam — 3g，q8h，120min infusion
  Arms: Meropenem and Pralurbactam
Drug: Saline — 100mL，q8h，60min infusion
  Arms: Meropenem and Pralurbactam
Drug: Ceftazidime-avibactam — 2.5g，q8h，120min infusion
  Arms: Ceftazidime-avibactam
Drug: Metronidazole — 0.915g，q8h，60min infusion
  Arms: Ceftazidime-avibactam

SUMMARY:
This is a Phase 3, randomized, double-blind, multicenter, positive control study to assess the efficacy, safety, and pharmacokinetics of Meropenem and Pralurbactam compared with Ceftazidime-avibactam in combination with Metronidazole in the treatment of adult complicated intra-abdominal infections (cIAI).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multicenter, positive control study to assess the efficacy, safety, and pharmacokinetics of Meropenem and Pralurbactam compared with Ceftazidime-avibactam in combination with Metronidazole in the treatment of adult complicated intra-abdominal infections (cIAI). Treatment duration for each cohort was 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 and ≤75 years of age.
* Diagnosed or highly suspected cIAI.
* Evidence of a systemic inflammatory response with at least one of the following:a. Fever ( temperature ≥ 38°C); b. hypotension (systolic blood pressure < 90 mmhg); c. abdominal pain; d. nausea and/or vomiting; e. physical examination found abdominal mass; f. mental state change; g. other circumstances.
* Female subjects must meet the following conditions: a. menopause for at least 1 year, or b. Sterilization has been performed, or C. Those who are fertile must meet the following conditions at the same time: the random pre-blood/urine pregnancy test is negative, effective contraceptive measures are taken during the study period and within 30 days after the last application of experimental drugs, and eggs are not donated, and they are not breastfeeding.
* Male subjects are willing to take effective contraceptive measures and not donate sperm during the study period and within 30 days after the last application of experimental drugs.
* Understand and abide by the research procedures and methods, voluntarily participate in this research, and sign an informed consent form .

Exclusion Criteria:

* Allergic to any carbapenem, cephalosporin, penicillin, metronidazole disodium phosphate, other beta-lactam drugs or other beta-lactamase inhibitors and their auxiliary materials.
* Non-complicated abdominal infection (infection is limited to abdominal organs), such as simple appendicitis and simple cholecystitis.
* Abdominal wall infection or abscess (infection has not spread into abdominal cavity).
* The creatinine clearance rate in the screening period is ≤50mL/min.
* The estimated survival time is less than 4 weeks.
* Those who have a history of drug abuse or drug abuse within 6 months before screening.
* Those who participated in other clinical trials within 28 days before randomization and used any test drugs or medical devices.
* Any physiological or psychological disease or condition that may increase the risk of the experiment, affect the compliance of the subject with the protocol or affect the completion of the experiment as judged by the researcher.
* Subjects are directly related persons who participated in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With a Clinical Response of "Cure" at the Test of Cure (TOC) Visit | Up to approximately 28 days
  Percentage of Participants With a Clinical Response of "Cure" at the Test of Cure (TOC) Visit

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Ju, MM, Study Chair — Qilu Pharmaceutical Co., Ltd.
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China